CLINICAL TRIAL: NCT04807608
Title: Study for the Evaluation of the Usability of EmbracePlus, Empatica Care Platform and Aura Algorithm
Brief Title: EmbracePlus, Care App and Aura Usability Study
Status: Completed | Type: Observational
Sponsor: Empatica, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2021-001
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Usability
Keywords: Usability; Wearable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Users: Each subject will be provided with a wearable device (smartwatch EmbracePlus manufactured by Empatica), to be worn every day outside of work hours for a total of 6 weeks. After the 6 weeks of data collection the participant will be asked to fill an online questionnaire related to the system usability (max 20 min).
  Interventions: Other: Usability Assessment

INTERVENTIONS:
Other: Usability Assessment — A survey will be administered to the subject at the end of the 6th week of product usage related to the wearable device and the related software platform's usability. Survey items will include both Likert-scale items that will be analyzed quantitatively and open-ended feedback that will be summarized qualitatively.

SUMMARY:
The purpose of this study is to evaluate the usability of the system which includes the wearable device, app and cloud data processing, including an algorithm (Aura) capable of detecting possible early signs of respiratory infections in healthy individuals.

In addition, the investigators would like to evaluate the presence of any allergic reactions to materials used in the manufacture of the EmbracePlus.

DETAILED DESCRIPTION:
The investigators wish to evaluate of the usability, according to the requirements of IEC 62366-1:2015/AMD 1:2020 of a wearable device - EmbracePlus, the Empatica Care app and Aura algorithm, an early-warning wearable/AI platform for alerting to COVID-19 and other possible respiratory infections before a person is symptomatic. The system consists is a smartwatch coupled with an AI algorithm (Aura) developed by Empatica. The Aura algorithm analyzes physiological signals and derived biomarkers (such as sleep patterns) in order to detect possible early signs of respiratory infection. It has been originally developed by Empatica, validated with influenza and rhinovirus data and is being currently validated for COVID-19 infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Participants must be between the ages of 18-99
2. Gender: No restrictions
3. Disease: healthy participants
4. Adult participant must either be able to give consent
5. Participants must be fluent in the language of the consent forms (Currently limited to English).
6. Participants must reside in the United States.
7. Participants should have a physical home address where they can receive the device
8. Participants must have a personal smartphone Apple or Android (at least iPhone 8 or Android 5.0)

Exclusion Criteria:

1. Participants must not have broken or injured skin at the wrist where EmbracePlus is worn, and they must be able to tolerate wearing EmbracePlus snugly for long periods of time. Thus, they should not have allergies to the material composition of the EmbracePlus smartwatch, or discomfort wearing a smartwatch during the night.
2. Participants are not willing to wear the device during nighttime
3. Participants should not have pre-existing cardiovascular disease or respiratory disease
4. Participants must not be pregnant or planning to become pregnant within two months at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women over 18, based in the US, without pre-existing pathologies that can affect their physiological parameters.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
EmbracePlus, Care App and Aura Usability: Based on user survey | After 6 weeks of system usage
  Determine the ease of use of the system composed of EmbracePlus, Care app and Aura algorithm and user satisfaction, by means of a survey items that include both Likert-scale items that will be analyzed quantitatively and open-ended feedback that will be summarized qualitatively.
EmbracePlus, Care App and Aura safety: total number (%) of AEs and SAEs | After 6 weeks of system usage
  The second primary endpoint will be the total number (%) of AEs and SAEs related to the device use

SECONDARY OUTCOMES:
EmbracePlus, Care app and Aura reliability with different smartphones | Single-point evaluation (baseline)
  Evaluate the reliability of the system with different brands and models of smartphone by means of participants reported bugs and problems

CONTACTS AND LOCATIONS:
Locations (1):
- Empatica Inc, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No